CLINICAL TRIAL: NCT06379581
Title: Photoacoustic Imaging for Three-dimensional Delineation of Skin Tumors
Brief Title: Skin Cancer Diagnostics Using Photoacoustic Imaging
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-04900-02
Record Dates: First submitted 2024-04-17; First posted 2024-04-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected skin tumors: With the help of photoacoustic imaging (PAI), determine the border between healthy tissue and tumor by determining the difference in chromophoric composition by their difference in absorption spectral features.

SUMMARY:
In this clinical study, photoacoustic imaging will be used on patients with suspected skin cancer (primarily melanoma, basal cell carcinoma, and squamous cell carcinoma) to determine the tumor borders both superficially and at a depth.

DETAILED DESCRIPTION:
The study will employ multispectral photoacoustic imaging in the spectral range between 680-970 nm to scan suspected skin tumors both in vivo and ex vivo. The hyperspectral data will then undergo rigorous spectral analysis with the objective to identify the spectral fingerprints associated with healthy tissue and tumor. Thereafter, a classification algorithm will be used to determine whether a pixel in the acquired image more likely identifies with healthy tissue or tumor, which is then repeated for all pixels in the images. As such, a 3D image can be reconstructed in which the tumor is visibly contrasted from healthy tissue. Achieving this goal will facilitate the diagnostic procedures and greatly reduce waiting times, clinical costs and potential patient suffering.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to perform surgical excision of lesion(s) suspected to be tumors.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled to perform surgical excision of lesion(s) at the Clinic of Dermatology, Lund, Skåne University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Tumor thickness | Enrollment is anticipated to last 1 year + final analyse 6 months
  Compare the estimated tumor thickness of tumor lesion with the provided thickness from the histopathological investigation.
Tumor size | Enrollment is anticipated to last 1 year + final analyse 6 months
  Compare the estimated tumor surface size of tumor lesion with the provided thickness from the histopathological investigation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthamology, Lund, Skåne University Hospital, Lund, Sweden